CLINICAL TRIAL: NCT05427487
Title: A Phase 1 Open-label, Non-randomized, Multi-cohort Clinical Study of Intratumoral IVX037 in Patients With Advanced or Metastatic Solid Tumours
Brief Title: Study of Intratumoral IVX037 in Patients With Advanced or Metastatic Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmVirx Pty Ltd (Industry)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-IVX001
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Gastric Cancer; Ovarian Cancer
Keywords: IVX037 virus sintilimab checkpoint gastric ovarian CRC
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Phase 1 open-label, non-randomized, multi-center clinical trial. The study is run in 2 parts. Part 1a is dose escalation of IVX037 monotherapy. Part 1b is IVX037 with checkpoint inhibitor, sintilimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1a (Experimental): IVX037 administered intratumorally, 1, 2 or 3 doses q2wks, Day 1, 15 and 29.
  Interventions: Biological: IVX037
- Part 1b (Experimental): IVX037 administered intratumorally 3 doses q2wks, for up to 7 doses. Sintilimab administration will commence on Study Day 8 and be administered every three weeks (Q3wks) at 200 mg/dose through to Study Day 344.
  Interventions: Biological: IVX037; Biological: Sintilimab

INTERVENTIONS:
Biological: IVX037 — Bioselected oncolytic RNA virus
Biological: Sintilimab — An immune checkpoint inhibitor
  Arms: Part 1b

SUMMARY:
This is a Phase 1 open-label, non-randomized, multi-center clinical trial of intratumoral IVX037 as monotherapy and in combination with an immune checkpoint inhibitor in patients with advanced micro satellite-stable (MSS) colorectal cancer, or gastric or ovarian cancer.

The study is run in 2 parts. Phase 1a is dose escalation IVX037 monotherapy and Phase 1b is IVX037 with checkpoint inhibitor, sintilimab.

DETAILED DESCRIPTION:
In Phase 1a, participants are treated with IVX037 alone by intratumoral administration as monotherapy. Participants will be enrolled by cohort, with a Safety Review Committee (SRC) reviewing any dose-limiting toxicities (DLTs) that develop within 21 days after the first, second, or third dose of IVX037 for Cohorts 1, 2 and 3, respectively. Cohorts in the dose escalation will consist of 3-6 participants.

Participants in Cohort 3 are permitted to receive up to seven doses of IVX037 in the absence of DLTs and at the discretion of the Investigator. The SRC will review Cohort 3 safety data once three participants have completed three doses of IVX037 and 21-days of safety data is available and will make a recommendation as to whether the dose expansion phase may commence.

In the dose expansion phase, up to 5 additional participants from each of the three tumor types will be enrolled and receive IVX037 at the MTD. A total of fifteen (15) participants (5 from each of the 3 tumor types) at the maximum tolerated dose will provide paired tumor biopsies, one taken on Day 1 prior to IVX037 intratumoral injection and a second one taken two weeks later on Day 15.

In Part 1b, a total of 45 participants (15 from each of the three tumor types) will be enrolled and receive the number of intratumoral doses of IVX037 that were deemed safe during Part 1a, in combination with an intravenous (IV) immune checkpoint inhibitor, sintilimab. Sintilimab administration will commence on Study Day 8 and be administered every three weeks (Q3wks) at 200 mg/dose through to Study Day 344.

ELIGIBILITY:
Inclusion Criteria:

1. Has either a histologically confirmed advanced colorectal, gastric/gastroesophageal adenocarcinoma, or ovarian cancer that has progressed or is not suitable for standard of care systemic therapies. Participants with colorectal cancer must have either a primary tumor or a biopsy of a metastatic tumor which has been shown to lack microsatellite instability (by PCR) or to have normal expression of mismatch repair enzymes (by immunohistochemistry). That is, a mismatch repair proficient mCRC tumor.
2. Progressed on or after at least one prior line of systemic therapy and must not have had more than 3 prior lines. Phase 1b only: participants with gastroesophageal cancer must have failed prior treatment with an immune checkpoint inhibitor.
3. Has at least one injectable tumor that meets RECIST1.1 criteria to be designated as a target lesion, and is:

   1. a liver lesion 1.0 to 6.5 cm (longest diameter) meeting RECIST criteria on baseline CT scan or MRI and suitable for injection under CT or ultrasound guidance, and participant has an estimated total tumor burden of disease < 1/3 of liver volume based on CT or MRI imaging, or
   2. A measurable lymph node, i.e., with a short axis diameter (SAD) of 1.5 cm to 6.5 cm, or
   3. Other solid tumor with a longitudinal diameter 1.0 cm to 6.5 cm.
   4. No other lesions (including non-injected lesions) greater than 6.5 cm (longest diameter).

   Note (i): Only 2 target lesions may be designated in any one organ but if an organ such as the liver has more than 2 lesions which can be injected, the others, up to 3 additional, may be designated as NTLs and injected. Alternatively, target and non-target lesions elsewhere up to a total of 5 may be selected for injection.

   Note (ii): Tumor lesions located in areas previously subjected to radiation or other locoregional therapies are not considered measurable unless there is a demonstrated progression in that lesion, as determined by the Investigator.
4. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
5. Has demonstrated adequate organ function defined in the protocol, from samples collected within 72 hours prior to the start of treatment.
6. Is a male or female from 18 to 85 years or age at the time of signing the informed consent.
7. Must be willing to abstain from activities or use proper birth control methods for the duration of the study:

   1. Female participants of child-bearing potential must be willing to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
   2. Male participants of child-bearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
8. The participant (or their legally acceptable representative if applicable) has provided written, informed consent prior to the initiation of any study procedures.
9. Female participants of child-bearing potential must have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
10. Participants must have fully recovered to NCI-CTCAE Grade 1 or better from AEs due to all previous anticancer therapies prior to entering this study. Note: Participants with Grade ≤ 2 AEs that are deemed not clinically significant by the Investigator may qualify for the study with approval by the Sponsor.
11. The participant has a life expectancy of greater than 6 months.

Exclusion Criteria:

Medical Conditions

1. The potential participant is deemed to be a candidate for hepatic surgery or locoregional therapy for liver lesions with curative intent or requires other systemic anti-cancer therapy.
2. The participant has clinically significant ascites (Grade ≥2).
3. Participants with any other concurrent uncontrolled illness, including mental illness or substance abuse, which may interfere with the ability of the participant to cooperate and participate in the trial; other examples of such conditions would include unstable or uncontrolled hypertension, unstable angina, myocardial infarction or cerebrovascular accident within 6 months of study entry.
4. The participant requires continuous systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 4 weeks prior to the first dose of study treatment. Single doses of corticosteroids for prophylaxis of allergic reactions during imaging studies with contrast are allowed within 4 weeks of study treatment.
5. The participant has not fully recovered from any effects of major surgery without significant detectable infection. Surgeries that require general anesthesia must have been completed at least 2 weeks before first dose of IVX037.
6. Participants with bleeding diathesis due to underlying medical conditions or the use of anticoagulation medications that is unable to be reversed by medical treatment.
7. Participants with tumors that lie close to an airway, major blood vessel or spinal cord, which, in the opinion of the Investigator, could cause occlusion, compression, or erosion of the vital structures.
8. Participants with multi-focal miliary disease without critical target lesions. Prior/Concomitant Therapy
9. Participants who have been previously treated with an immune checkpoint inhibitor (e.g., an anti-CTLA-4, anti-PD-1 or anti-PD-L1) must have completed their last dose at least 28 days prior to Day 1 and have demonstrated progressive disease during or following the immune checkpoint inhibitor therapy. The participant must also have no medical history of immune mediated adverse events including infusion (hypersensitivity) reactions ≥ Grade 3 (CTCAE), with the exceptions of adequately treated hypothyroidism and type 1 diabetes mellitus (hyperglycemia) resulting from past treatment with an immune checkpoint inhibitor and non-exfoliative dermatologic reactions such as vitiligo. A history of Grade 2 immune-mediated infusion reactions to an immune checkpoint inhibitor while receiving adequate prophylactic treatment for hypersensitivity reactions is also exclusionary.
10. Participants who require prohibited treatments (i.e., non-protocol-specified anticancer pharmacotherapy, surgery, or radiotherapy for treatment of malignancy). Prohibited medications must be ceased at least 21 days or 5 half-lives (whichever is longer) prior to Day 1.

    Prior/Concurrent Clinical Study Experience
11. Is currently participating and receiving other study therapy including an investigational agent or device within 4 weeks of Day 1.
12. Participants who have received a live vaccine within 4 weeks of the first day of planned IVX037 treatment or any other vaccine including killed virus and mRNA vaccines within 2 weeks of the first day of planned IVX037 treatment.

    Diagnostic Assessments
13. Participant with active (i.e., symptomatic or growing) central nervous system (CNS) metastases. Participants with CNS metastases are eligible for the trial if the metastases have been treated by surgery and/or radiotherapy, the participant is off corticosteroids for at least 2 weeks prior to first dose of IVX037 and have stable disease on imaging for 3 months prior to Day 1.
14. Participant has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by the local health authority.
15. Participant has a severe infection or other uncontrolled active infectious disease requiring treatment that would interfere with the evaluation of safety and efficacy or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.
16. Has a history of other malignancies within the previous 3 years, except for locally curable cancers which have been apparently cured such as basal cell or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast or other cancers with low risk of recurrence in discussion with the Sponsor.
17. Has a history of drug-induced interstitial lung disease or non-infectious pneumonitis requiring steroids, except for those induced by radiation therapies.
18. Has a history of a prior organ transplantation, including allogenic stem-cell transplantation.
19. Has an active or known documented autoimmune disease within the past 2 years that has required systemic treatment.
20. Has a history of primary immunodeficiency.
21. Has an evidence of small bowel obstruction as determined by air/fluid levels on computed tomography (CT) scan, or recent hospitalization for small bowel obstruction within 3 months prior to starting trial treatment.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.

    Other Exclusions
23. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the Screening visit through 120 days after the last dose of trial treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a - feasibility, safety, and tolerability of intratumoral IVX037 when administered to patients with advanced colorectal, ovarian or gastric cancers | 21 days after following cessation of study intervention
  Incidence of dose-limiting toxicities (DLTs), viral excretion, adverse events (AEs), serious adverse events (SAEs) and changes from baseline in clinical chemistry and hematology laboratory values. Safety overall will be measured by CTCAE v5.
Phase 1b - safety and efficacy of intratumoral IVX037 in combination with an intravenous immune checkpoint inhibitor | 21 days after following cessation of study intervention
  Viral excretion, incidence and severity of AEs, SAEs, and changes from baseline in clinical chemistry and hematology laboratory values. Efficacy will be assessed through iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Shafren, Study Chair — ImmVirx Pty Ltd; Oksana Zdanska, Study Director — ImmVirx Pty Ltd
Locations (3):
- Australia (3):
  - Sydney site, Sydney, New South Wales
  - South Australia site, Adelaide, South Australia
  - Melbourne Site, Melbourne, Victoria

REFERENCES:
- [Result] Liu J., Tebbutt, N., Price, T., Hus, E., Al-Asady, R., Shafren, D., Zdanska, O., Croll, N., Wong, M. Phase 1a/b open-label, non-randomized, multi-centre clinical trial of intratumoral IVX037 alone and in combination with anti-PD1 in patients with advanced microsatellite stable (MSS) colorectal, gastroesophageal or ovarian cancer: trial in progress. Medical Oncology Group of Australia (MOGA) Sydney, Australia Conference Poster 2024
- [Result] Liu, J., Price, T., Tebbutt, N., Hsu, E., Al-Asady, R., Shafren, D., Croll, N., Wong, M. Phase 1a open-label, non-randomized, multi-center clinical trial of intratumoral IVX037 in patients with advanced microsatellite stable (MSS) colorectal, gastroesophageal or ovarian cancer. SITC 2023 Poster Presentation. Abstract Number 649